CLINICAL TRIAL: NCT02885584
Title: Conventional Mechanical Ventilation and High Frequency Percussive Ventilation: Comparison of Their Effects on Alveolar Recruitment and Distension by CT-scan in Early ARDS Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2013-11; 2013-A00465-40 (Other: Ansm)
Record Dates: First submitted 2016-08-26; First posted 2016-08-31 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: ARDS
Keywords: Mechanical ventilation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transpulmonary pressure controlled mechanical ventilation (Experimental): transpulmonary pressure will be used for ventilation settings
  Interventions: Device: High frequency percussive ventilation
- Conventional pressure-controlled mechanical ventilation (No Intervention): transpulmonary pressure will not be used for ventilation settings

INTERVENTIONS:
Device: High frequency percussive ventilation
  Arms: Transpulmonary pressure controlled mechanical ventilation

SUMMARY:
High frequency percussive ventilation (HFPV) is a high frequency ventilation mode in which high frequency pulses accumulate to generate a low frequency tidal volume at a controlled airway pressure. Previous studies have suggested a protective effect of HFPV on lung injury. The goal of our study is to compare, in early ARDS patients, the effects of conventional mechanical ventilation and of high frequency percussive ventilation on alveolar recruitment and distension evaluated by CT-scan

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing invasive ventilation for more than 24h
* ARDS patient

Exclusion Criteria:

* Pneumothorax drained or not
* Patient undergoing extracorporel mechanical oxygenation
* Patient who had a pneumonectomy partiel or total

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-12; Primary Completion 2016-05 (Actual); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Percent of patients exhibiting under HFPV an increase of at least 15% of normally aerated end-expiratory lung volume | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique-Hôpitaux de Marseille; Antoine ROCH, MD/PhD, Principal Investigator — Assistance Publique-Hôpitaux de Marseille
Locations (1):
- Assistance Publique-Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No